CLINICAL TRIAL: NCT04422015
Title: Unravelling Disease Tolerance and Host Resistance in Afebrile P. Falciparum Infections: a Prospective Study in Mozambican Adults
Brief Title: Biological Mechanisms in Afebrile P. Falciparum Malaria
Acronym: AsintMal
Status: Completed | Type: Observational
Sponsor: Alfredo Mayor (Other)
Collaborators: Centro de Investigação em Saúde de Manhiça (Other); Stanford University (Other); University of Florida (Other)
Responsible Party: Sponsor-Investigator, Alfredo Mayor, Associate Research Professor, Barcelona Institute for Global Health
Organization: Barcelona Institute for Global Health (Other)
Other Study IDs: 1R01AI150521 (NIH)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Falciparum Malaria
Keywords: afebrile; resistance; tolerance
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This project aims to disentangle the role of host immune resistance and disease tolerance in afebrile malaria infections, with the goal of guiding context-adapted tactics to target this hidden reservoir, as well as to develop new approaches to clear malaria infection and reduce its severity through host-directed therapies.

DETAILED DESCRIPTION:
Asymptomatic Plasmodium falciparum (Pf) infections debilitate the health of affected population while representing a hidden source of parasite transmission that can compromise elimination efforts. The lack of consensus on the best strategy to deal with this asymptomatic reservoir is partly due to the poor knowledge on the biological mechanisms underlying these subclinical infections. Preliminary results in Mozambique show that afebrile adults with a Pf infection detected by rapid diagnostic tests can progress to fever (10%), clear the infection (20%) and stabilize at low-density (50%) or high-density (20%) parasitemias. The study hypothesis is that these four main trajectories are driven by antibodies against Pf variant antigens, codified by the var gene family and expressed on the surface of infected erythrocytes, which would clear the infection unless the parasites develop immune evasion mechanisms, and by tolerance factors that minimize parasite-induced pathology and sustains host homeostasis.With the overarching goal of identifying key biological factors sustaining afebrile malaria infections, this project will establish a cohort of afebrile Mozambican adults followed during one month to identify subjects who can reduce pathogen load and eventually clear the infection, those who maintain infections at high-density and afebrile levels (tolerant), and those who fail to establish disease tolerance and progress to fever. Circulating and overall parasite biomass will be quantified, and new infections will be identified during follow-up using next-generation sequencing. Clinical samples from individuals with low and high parasite densities will be used to test whether parasitological trajectories of afebrile Pf infections correlate with host antibody immunity against erythrocyte surface antigens and the transcription of Pf var genes involved in cytoadhesion and immune evasion. Cytometry by time of flight and global mass spectrometry will be applied on clinical samples from afebrile individuals with high parasite densities (tolerant) and those progressing to fever (non-tolerant) to identify leukocyte populations and metabolic pathways involved in the regulation of inflammation, tissue damage and normoglycemia that support host-parasite relationships at afebrile levels. The expected outcome of this project is the identification of key molecular drivers of afebrile Pf infections for a better understanding of the relevance of these infections in different transmission setting which may require context-specific control approaches, as well as for the development of new tools to achieve sterilizing immunity and enhance disease tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤60 years
* A positive RDT and microscopy for P. falciparum
* Axillary temperature < 37.5ºC without history of fever during the last 24h
* No danger signals for severe malaria (Impaired consciousness, respiratory distress, multiple convulsions, prostration, shock, abnormal bleeding, jaundice)
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Signed informed consent after explaining the purpose of the study

Exclusion Criteria:

* Age <18 years or >60 years
* Axillary temperature ≥37.5ºC
* Reported pregnancy
* Presence of any sign/symptom of malaria (Vomiting, diarrhea, weakness, dizziness, fainting, itching, urticarial)
* Presence of any other co-existing clinical condition that would not allow the individual to be considered a "healthy" afebrile carrier
* Having received antimalarial medication in the preceding 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals (temperature below 37.5ºC) with a P. falciprum infection confirmed by RDT and microscopy
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals developing fever | 1 month
  Development of axilary temperature higher or equal than 37.5ºC

SECONDARY OUTCOMES:
Proportion of individuals clearing the infection | 1 month
  Clearance of parasite infection as detected by qPCR
Proportion of individuals maintaining infections without fever | 1 month
  Confirmed P. falciparum ifection at day 28 by qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Fundação Manhiça/Manhiça Health Research Center, Manhiça, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided